CLINICAL TRIAL: NCT01254201
Title: The Pathogenesis of Idiopathic Dry Eyes
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Roni Shtein, Assistant Professor of Ophthalmology and Visual Sciences, University of Michigan
Other Study IDs: HUM00013091
Record Dates: First submitted 2010-12-03; First posted 2010-12-06 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Dry Eye; Fibromyalgia
MeSH Terms: conditions — Dry Eye Syndromes; Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Dry Eye: Female patients over the age of 18 years with ocular complaints of dryness, grittiness, irritation, or related symptoms, without any identifiable cause.
- Fibromyalgia: Female patients over the age of 18 years diagnosed with Fibromyalgia.
- Healthy Control: Female patients over the age of 18 years with no symptoms of dry eyes and with no known diagnosis of Fibromyalgia.

SUMMARY:
Dry eyes are a very common complaint. In some patients, we can identify the reason for the dryness; however, in others the dryness has no clear cause. Dryness can lead to eye irritation, redness, and sometimes changes in vision. Fibromyalgia is a condition of chronic pain that is poorly understood but seems to have a component of altered sensory processing. People with fibromyalgia tend to complain of dry and irritated eyes at a higher rate than the general population. We plan to evaluate patients with dry eye symptoms for abnormalities in sensory processing and in their autonomic nervous system. We hope to learn about possible relationships between dry eye symptoms and fibromyalgia in order to better understand and treat these conditions.

DETAILED DESCRIPTION:
Dry eye and fibromyalgia syndromes are most prevalent in women. Therefore, female patients seen in Kellogg Eye Center for ocular complaints of dryness, grittiness, irritation, or related symptoms, without any identifiable cause, will be offered enrollment into the study. These individuals will be compared to both a "positive control" group (fibromyalgia patients) and a healthy control group. We hypothesize that the patients seen with irritative symptoms will have autonomic and sensory processing profiles similar to fibromyalgia patients, and both groups will differ from healthy controls. All study participants will have an extensive ophthalmological exam in addition to autonomic and sensory testing, in order to more fully characterize the underlying mechanism(s) of these symptoms.

Recruitment:

Female patients over the age of 18 with the above mentioned complaints will be told of the study at the time of their visit. They will be given a copy of the study consent form to take home with them or one will be mailed to them. Additionally, from CareWeb billing records, or from other University of Michigan Ophthalmologists, a list of patients who have previously been seen (within the last year) in the Ophthalmology Comprehensive Clinic for dry eyes complaints will be identified and contacted by US mail with a recruitment letter uploaded. If the patient is interested, the letter will list research staff contact information, who patients may then contact. If the patient does not contact research staff by phone or email, research staff may follow-up the letter by phone no earlier than one week after it is mailed. If patients are not interested, a phone number will be listed allowing patients to opt-out of being contacted about the study by phone in the future. Follow-up phone calls will utilize a phone script.

Patients who are interested in participating will be contacted by the study coordinator for further discussion to see if they meet the inclusion and exclusion criteria and to schedule a visit to the Cornea Clinic for an ophthalmic evaluation. At the time of this visit, patients will be asked to sign the consent form and be given a study identification number that will be used exclusively in patient identification in study materials. These patients will then be scheduled to be seen at the Chronic Pain and Fatigue Research Center at Dominos Farms for the remaining sensory and autonomic testing. All patient study information will be collected and encoded according to HIPAA guidelines and institutional review board approval. The plan is to enroll 50 patients into Group 1 over a 12 month enrollment period.

The study group will be compared to two groups of age matched patients, 25 with known FM (Group 2) and 25 healthy controls (Group 3). These patients will be identified by searching the patient registry that includes more than 400 FM and healthy control patients who have already undergone the standardized sensory and autonomic evaluations at the Chronic Pain and Fatigue Research Center. The study coordinator will then contact the individuals that are identified in the registry that meet these criteria, and they will be asked if they are interested in enrolling in this particular study (all individuals in the registry have given consent to be contacted for additional studies for which they are eligible). FM patients and controls who agree to participate will be asked to sign the consent form and be scheduled for the ophthalmic evaluation at the Cornea Clinic.

Ophthalmic Evaluation:

Individuals in all three groups will be seen in the Cornea Clinic at the Kellogg Eye Center and will receive a complete ophthalmic evaluation including the following objective measures of ocular and visual sensation:

* Visual acuity will be assessed in each eye separately, using a Snellen acuity chart for distance and a Jaegar reading card for near vision. Additional notations will be made for subjective evaluation of patient's level of satisfaction with corrected acuity during testing.
* Shirmer's testing with anesthesia will be performed on all patients. This test involves the use of small strips of filter paper placed in the lower eyelids after instillation of anesthetic eyedrops for the assessment of tear production.
* Corneal fluorescein and conjunctival lissamine green staining patterns will be assessed as a measure of ocular surface integrity. Staining will be measured using the Oxford grading scale from 0 (no staining) to 5 (severe staining)
* Tear break up time is evaluated while fluorescein stain is still in the eye. The patient is instructed not to blink and the tear film is observed through the slit lamp. If the smooth layer tear film begins to visibly break up prior to 10 seconds, the patient's tear film is considered abnormal.
* Ocular complaints will be quantified with the use of the Ocular Surface Disease Index Questionnaire - a validated 15 question survey that evaluates dry eye symptoms as well as the National Eye Institute Visual Functioning Questionnaire - a validated 25 question survey that evaluates overall visual function.
* Accommodation, or the ability to shift visual focus from distance to near, will be measured with the Marco auto-refractor separately for each eye. Accommodation is a physiologic measure of the eye's ability to shift focus and naturally decreases with age.
* Central corneal sensation will be measured using Cochet-Bonnet esthesiometry. The esthesiometer is an instrument that comprises a slender nylon filament that is retracted in 0.5 cm increments until the filament is sensed on the cornea.
* Confocal Microscopy - The patients' eyes will be viewed using a high power microscope to carefully evaluate the corneal nerve layer. This microscope looks at the layers of the cornea (or window) of the eye. After numbing drops are placed in eye, a gel to lubricate will also be placed in the eye. The microscope comes into close proximity to the eye. The patient will feel the microscope against his/her eyelashes while looking at a red light. Three scans providing a clear view of the sub-epithelial corneal nerve layer will be performed on each patient.

Sensory and Autonomic Evaluation:

Patients seen in the Chronic Pain and Fatigue Research Center at Dominos Farms will be evaluated by several modalities for measures of altered sensory processing and autonomic dysfunction:

* Questionnaires of demographic and disease status information will be collected using a general form that includes age, sex, race, marital status, education level, ethnicity, chronicity of pain, believed cause of pain, and events associated with the onset of pain. Participants will also complete a battery of self-report questionnaires that characterize their functional status, pain and fatigue symptoms, cognitive difficulties, affective status, pain beliefs, perceived stress, perceived social support, coping strategies, sleep quality, and history of abuse. The questionnaire battery takes approximately 1 hour to complete.
* Pressure pain sensitivity is assessed at the thumbnail using a hydraulic device that consists of a plastic housing and piston driving a hard rubber 1 cm2 probe. After positioning the device on the left thumb, subjects will receive an ascending series of discrete 3 second-duration pressure stimuli beginning at 0.5 kg and increasing in 0.5 kg steps to a maximum of 10 kg (or subjective maximum less than 10 kg). Subjects will rate the intensity of the evoked sensations using the sensory intensity Box scale, a combined analog descriptor scale that superimposes verbal descriptors, spaced according to ratio-scale values, on a 0-20 graphical numerical category scale.22,23 The pain testing session lasts about 45 minutes.
* Tender point assessment: a standard means of confirming the diagnosis of fibromyalgia. During this assessment, the examiner will use their thumb to apply minimal pressure on pre-designated body points (such as the base of the neck, or back of the arm) and ask if the patient is sensitive or 'tender' at these various points. Most individuals do not describe this assessment as painful.
* Auditory sensitivity testing involves a hearing screening performed according to the American Speech-Language-Hearing Association guidelines.24 This includes a brief case history, otoscopic inspection, and a 25 dB HL pure-tone screen at 1000, 2000 and 4000 Hz and 35 dB HL at 500 Hz. This testing is to assure that there are no hearing abnormalities that would cause abnormalities on the research test of interest, the Judgment of Loudness Discomfort Levels (LDLs). This testing is performed using pure tone acoustic stimuli at an octave frequency of 2000 Hz and signal range from 40 to 100 dB. The patient is instructed to indicate a rating of discomfort for each volume at which the acoustic signal is presented. This test will be performed in both ascending step-wise and random order patterns, and takes approximately 45 minutes. Each patient will also complete a hyperacusis questionnaire,25 through which they will indicate their experiences of real-life auditory sensitivity.
* Dysautonomia will be assessed centrally by monitoring variations in heart rate. Heart rate variability information is obtained by use of a Holter monitor. Individuals will remain supine for the first 5 minutes of the examination. For the remaining time period (total: approximately 60 minutes), the Holter monitor will record a continuous electrocardiogram (ECG) of the heart's electrical activity in response to varying but standardized study related tasks such as questionnaire completion, discussions with study personnel, and listening to instructions. Frequency domain analysis using fast Fourier transformations yields information about the amount of the variance (power) in the heart's rhythm explained by periodic oscillations of the heart rate at various bands, including the high, low, and very low frequencies.26 Fluctuations over time in the interval between normal heartbeats is recorded and quantified by analysis of variability between beats.

ELIGIBILITY:
Inclusion Criteria:

Healthy Controls:

Female over the age of 18, No symptoms of dry eyes, Must be able to read text on the computer screen and understand English, and not have a physical impairment that prevents you from completing a paper and pencil questionnaire or using a tablet computer

Fibromyalgia:

Female over the age of 18, No symptoms of dry eyes, Been diagnosed with fibromyalgia, Must be able to read text on the computer screen and understand English, and not have a physical impairment that prevents you from completing a paper and pencil questionnaire or using a tablet computer

Dry Eye:

Female over the age of 18, have symptoms of dry eyes, Must be able to read text on the computer screen and understand English, and not have a physical impairment that prevents you from completing a paper and pencil questionnaire or using a tablet computer

Exclusion Criteria:

Pregnant or breast feeding, use of medicated eye drops in last month (Artificial tears ok), diagnosis of autoimmune or rheumatologic disease (e.g. rheumatoid arthritis, crohn's disease, lupus, multiple sclerosis, etc), heart condition requiring daily medications (e.g. angina, congestive heart failure), COPD or asthma requiring daily inhalers (rescue inhalers ok), history of cancer in the past 2 years (skin cancer is ok), use of oral antihistamine medications (e.g. benadryl, claritin, clarinex, zyrtec, allegra, etc), use of oral anticholinergic medications (e.g. scopolamine, ditropan, detrol, ipratropium, etc)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Females aged 18 yrs or older in the community or seen in Kellogg Eye Center will be offered enrollment into the study.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2008-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roni Shtein, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Kellogg Eye Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No